CLINICAL TRIAL: NCT04304313
Title: A Pilot Study of Sildenafi in the Treatment of COVID-19
Brief Title: A Pilot Study of Sildenafil in COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GST-G1
Record Dates: First submitted 2020-02-14; First posted 2020-03-11 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sildenafil citrate tablets (Experimental)
  Interventions: Drug: Sildenafil citrate tablets

INTERVENTIONS:
Drug: Sildenafil citrate tablets — 0.1g/day for 14 days

SUMMARY:
Observe the efficacy and safety of G1(Sildenafil citrate tablets) in patients with COVID-19 under clinical actual diagnosis and treatment conditions

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as COVID-19:

   1. mild patient: fever,respiratory and other symptoms, the manifestation of pneumonia can be seen on imaging.
   2. severe patients: meet the definition of severe pneumonia(comply with any of the followings): Shortness of breath,RR≥30 bpm;In a resting state:SPO2≤93%;PaO2/FiO2≤300mmHg.
2. Age≥18 years old,unlimited gender.
3. Patients who cannot stop the following drugs during the trial:erythromycin or strong inhibitors of CYP3A4 (such as saquinavir,ketoconazole,itraconazole),nonspecific inhibitors of CYP (such as cimetidine),HIV protease inhibitors (such as ritonavir).
4. Willing to participate in this study,signed Informed Consent and willing to participate in regular follow-up during the study.

Exclusion Criteria:

1. Suffer from severe cognitive impairment or mental illness.
2. Pregnant and lactating women.
3. Patients taking nitric oxide drugs and nitrates in any dosage form.
4. Patients with malignant tumors;AMI, stroke or life-threatening arrhythmias within 6 months;hereditary pigmented retinitis;heart failure or unstable angina pectoris of coronary heart disease;patients with severe hypotension and hypertension.
5. Patients who are allergic to the study drug or the researcher believes it is not appropriate.
6. Participate in other clinical studies at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-02-09 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-11-09 (Estimated)

PRIMARY OUTCOMES:
Rate of disease remission | 14 days
  1. fever,cough and other symptoms relieved with improved lung CT;
  2. SPO2>93% or PaO2/FiO2 >300mmHg without oxygen inhalation.
Rate of entering the critical stage | 14 days
  Comply with any of the followings:
  1. Respiratory failure occurs and requires mechanical ventilation;
  2. Shock;
  3. Patients combined with other organ failure need ICU monitoring and treatment.
Time of entering the critical stage | 14 days
  Comply with any of the followings:
  1. Respiratory failure occurs and requires mechanical ventilation;
  2. Shock;
  3. Patients combined with other organ failure need ICU monitoring and treatment.

SECONDARY OUTCOMES:
Rate of no fever | 14 days
Rate of respiratory symptom remission | 14 days
Rate of lung imaging recovery | 14 days
Rate of C-reactive protein (CRP) recovery | 14 days
Rate of Biochemical criterion (CK, ALT, Mb) recovery | 14 days
Rate of undetectable viral RNA (continuous twice) | 14 days
Time for hospitalization | 14 days
  From the date of enrollment to the time when the subject is released from the hospital or transferred to the corresponding department for treatment of other diseases according to the condition.
Rate of adverse event | 14 days
  All adverse events will be coded and described using the International Medical Terms Dictionary (MedDRA).

CONTACTS AND LOCATIONS:
Locations (1):
- Department and Institute of Infectious Disease, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sultana J, Crisafulli S, Gabbay F, Lynn E, Shakir S, Trifiro G. Challenges for Drug Repurposing in the COVID-19 Pandemic Era. Front Pharmacol. 2020 Nov 6;11:588654. doi: 10.3389/fphar.2020.588654. eCollection 2020. PMID 33240091